CLINICAL TRIAL: NCT00206687
Title: Study of the Safety, Tolerability and Efficacy of Spheramine Implanted Bilaterally Into the Postcommissural Putamen of Patients With Advanced Parkinson's Disease
Brief Title: STEPS Trial - Spheramine Safety and Efficacy Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was completed, only life long extended follow-up phase was discontinued after 12 years.
Sponsor: Bayer (Industry)
Collaborators: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91039; 305405 (Other: Company Internal); NCT00059007 (obsolete NCT alias); NCT00185406 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: Spheramine (BAY86-5280)
- Arm 2 (Sham Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Biological: Spheramine (BAY86-5280) — Bilateral implantation of Spheramine into the postcommissural putamen, each side at a dose of 325,000 cells
  Arms: Arm 1
Procedure: Placebo — Sham surgery procedure without penetration of the dura mater. Nothing wil be implanted into the brain.
  Arms: Arm 2

SUMMARY:
The purpose of the study is to explore the safety, tolerability and efficacy of Spheramine (cultured human retinal pigment epithelial cells on microcarriers) in Parkinson's Disease patients with advanced disease who have insufficient symptom control by optimum oral medication. Patients are randomized to receive Spheramine injections into both hemispheres or a sham surgical procedure in a ratio of 1:1. A three month pretreatment period must be completed prior to surgery. Time to endpoint is 24 months.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. and Schering AG, Germany.Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc., Schering AG Germany has been renamed to Bayer Schering Pharma AG, Germany. Bayer HealthCare Pharmaceuticals, Inc.and Bayer Schering Pharma AG, Germany are the sponsors of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Parkinson's disease for at least 5 years
* Good response to L-dopa
* Age 30 to 70 years
* Optimum oral therapy

Exclusion Criteria:

* Tremor only
* Dementia
* Very severe dyskinesia
* Previous brain surgery including deep brain stimulation
* Malignant disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-01-08 (Actual); Primary Completion 2012-05-14 (Actual); Study Completion 2012-05-14 (Actual)

PRIMARY OUTCOMES:
Change in UPDRS part III (Motor Score) in the defined medication at 12 months post surgery | 12 months post surgery

SECONDARY OUTCOMES:
Change in total UPDRS in ON and OFF at 12 months post surgery | 12 months post surgery
Change in UPDRS Part III in ON at 12 months post surgery | 12 months post surgery
Amount of L-dopa reduction at 12 months post surgery | 12 months post surgery
Activities of Daily Living subscore of the UPDRS at 12 months post surgery | 12 months post surgery
Quality of Life as assessed by PDQ-39, SF-36 and EQ-5D at 12 months post surgery | 12 months post surgery
Percent time spent in ON and OFF at 12 months post surgery | 12 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (15):
- United States (10):
  - Birmingham, Alabama
  - Los Angeles, California
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - New York, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Germany (4):
  - Marburg, Hesse
  - Homburg, Saarland
  - Dresden, Saxony
  - Hamburg
- Barcelona, Spain

REFERENCES:
- [Derived] Gross RE, Watts RL, Hauser RA, Bakay RA, Reichmann H, von Kummer R, Ondo WG, Reissig E, Eisner W, Steiner-Schulze H, Siedentop H, Fichte K, Hong W, Cornfeldt M, Beebe K, Sandbrink R; Spheramine Investigational Group. Intrastriatal transplantation of microcarrier-bound human retinal pigment epithelial cells versus sham surgery in patients with advanced Parkinson's disease: a double-blind, randomised, controlled trial. Lancet Neurol. 2011 Jun;10(6):509-19. doi: 10.1016/S1474-4422(11)70097-7. Epub 2011 May 10. PMID 21565557